CLINICAL TRIAL: NCT04051931
Title: The Copmparison of Accuracy of PtcCO2 and in PetCO2 in COPD Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shanshan Zha, doctor, The First Affiliated Hospital of Guangzhou Medical University
Other Study IDs: 2019-27
Record Dates: First submitted 2019-07-29; First posted 2019-08-09 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- stable COPD group: include COPD patients with stable state
- AECOPD group: include COPD patients with acute exacerbation

SUMMARY:
The pathophysiological characteristics of COPD is irreversible airflow restriction which may influence the gas exchange and cause the abnormal PaO2 and PaCO2. Assessment of the partial arterial pressure of carbon dioxide (PaCO2 ) is the 'gold standard' for the evaluation of the adequacy of alveolar ventilation.Method used mostly nowadays : arterial puncture which is accurate but is invasive 、painful、 non-dynamic and there is risk of infection and tissue、nerve damage. Noninvasive measurement methods (Most commonly used)： end-tidal CO2（ ETCO2）、 transcutaneous CO2(TcCO2). They all can monitor the PaCO2 dynamically、 noninvasively, but is existence of controversy of the accuracy. So the investigators want to compare the accuracy of these two noninvasive methods for assessment of PaCO2.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients

Exclusion Criteria:

* hemodynamics is unstable;
* any other lung disease despite COPD；
* other diseases influencing experiments: Cognitive impairment disease、 mouth and nose trauma.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stable and acute axcerbation COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
concordance between the values of PetCO2 and PaCO2 measured at the same time | 1 hour
  concordance between the values of PetCO2 and PaCO2 measured at the same time
concordance between the values of PtcO2 and PaCO2 measured at the same time | 1 hour
  concordance between the values of PtcO2 and PaCO2 measured at the same time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zha S, He Z, Niu J, Huang Q, Liang Z, Zhou Z, Yang H, Lin S, Guan L, Zhou L, Chen R. Comparison of prolonged exhalation end-tidal CO(2) and transcutaneous CO(2) monitoring in COPD patients. Crit Care. 2026 Jan 20. doi: 10.1186/s13054-025-05834-5. Online ahead of print. PMID 41559738